CLINICAL TRIAL: NCT06089252
Title: Efficacy of Lazolex® Gel in the Treatment of Herpes Simplex Mucocutaneous Infections and the Prevention of Recurrences: A Pilot Study
Brief Title: Efficacy of Lazolex® Gel in the Treatment of Herpes Simplex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iveriapharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-000032
Record Dates: First submitted 2023-09-27; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: HSV Infection
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Intervention Model Description: Lazolex gel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSV-1, HSV-2 (Other): All participants were assigned to receive topical treatment with Lazolex® Gel. Patients were given the gel at the end of the screening visit (day 0) by the attending physicians.,e gel was applied to the lesion four times a day over a 10-day period, with the Lrst application at 9 am and the fourth at 9 pm. Patients administered Lazolex® Gel to the a2ected areas themselves.
  Interventions: Drug: walnut extract

INTERVENTIONS:
Drug: walnut extract — Four times a day over a 10-day period
  Other Names: Lazolex gel

SUMMARY:
Study aimed to evaluate the efficacy and tolerance of Lazolex®, an emollient gel, to treat mucocutaneous lesions caused by herpes simplex virus.

DETAILED DESCRIPTION:
A single-center, single-arm, open-label, phase II clinical trial was conducted with 30 patients divided into two groups: 15 patients with herpes simplex virus type 1 (HSV-1) infections and 15 with herpes simplex virus type 2 (HSV-2) infections. All received topical treatment with Lazolex® Gel four times daily for 10 days. The efficacy and tolerance of the treatment were evaluated on day 10 and day 20 after the study started. In addition, recurrence rates were evaluated before treatment with Lazolex® and after a 4-year follow-up period after treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute or chronic herpes simplex mucocutaneous infection,
* mild course of disease (defined as body temperature <37.2°C and without signs of general infirmity),
* application of last treatment for herpes simplex infection >3 months,
* available to cooperate during the study,
* provision of written informed consent.

Exclusion Criteria:

* abnormal laboratory results,
* hypersensitivity to the product or its components,
* pregnancy or breastfeeding,
* acute/ chronic renal or liver failure,
* history of migraine,
* organic brain lesion,
* generalized anxiety disorder,
* blood supply disturbance in the vertebrobasilar pool,
* stage 3 essential hypertension,
* concomitant acute or decompensated disease that could affect the study results,
* intake of acyclovir, antibiotics, immunosuppressants, antimetabolites, or glucocorticosteroids during 3-month period prior to the study,
* concomitant participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11-27 (Actual); Primary Completion 2007-12-28 (Actual); Study Completion 2008-01-28 (Actual)

PRIMARY OUTCOMES:
Course of the disease | 10 days
  Lazolex® Gel was classified as effective if herpes lesions improved or healed after treatment. The median effective time (ET50), defined as the time (in days) needed to reach complete recovery in 50% of the patients, was used as the main variable for Lazolex® Gel efficacy.
Change in outbreak frequency | 10 days
  Lazolex® Gel was classified as effective if herpes lesions improved or healed after treatment. The median effective time (ET50), defined as the time (in days) needed to reach complete recovery in 50% of the patients, was used as the main variable for Lazolex® Gel efficacy.
Change in outbreak frequency | 4 years
  Change in outbreaks along time

SECONDARY OUTCOMES:
The degree of patient satisfaction | 10 days
  The level of patient satisfaction with treatment efficacy was categorized as high, medium, or low using a self-questionnaire.
Number of complaints and symptoms | 10 days
  Tolerance outcomes were evaluated using both objective and subjective criteria. The objective criteria included the comparison of laboratory tests and physical examinations before and after Lazolex® Gel treatment. The subjective criteria included complaints and symptoms reported by patients. In the event of adverse reactions, they were assessed by attending physicians. Individual tolerance was categorized as follows:
  Very satisfactory: No clinically significant changes in physical examination or laboratory tests, and no adverse reactions.
  Satisfactory: Insignificant changes in physical examination or laboratory tests, or mild adverse reactions that do not require a change in treatment.
  Unsatisfactory: Significant changes in physical examination or laboratory tests and/or the occurrence of adverse reactions that require the withdrawal of the product, as well as prescribing treatment to address the adverse reaction

CONTACTS AND LOCATIONS:
Overall Officials: Tina A. Kituashvili, Ph.D,, Principal Investigator — National Center of Dermatology and Venereology, Tblisi (Georgia)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kituashvili TA, Kvirkvelia VG, Galdava GG, Archvadze NG. Efficacy of Lazolex(R) Gel in the Treatment of Herpes Simplex Mucocutaneous Infections and the Prevention of Recurrences: A Pilot Study. Can J Infect Dis Med Microbiol. 2022 Nov 16;2022:4413679. doi: 10.1155/2022/4413679. eCollection 2022. PMID 36437891
- See also: Can J Infect Dis Med Microbiol — https://www.ncbi.nlm.nih.gov/